CLINICAL TRIAL: NCT05229939
Title: Performances of Estimated Glomerular Filtration Rate Equations in Kidney Transplant Recipients
Brief Title: Estimating Glomerular Filtration Rate in Kidney Transplant Recipients
Status: Completed | Type: Observational
Sponsor: Paris Translational Research Center for Organ Transplantation (Other)
Responsible Party: Sponsor
Other Study IDs: KRSeGFR2021
Record Dates: First submitted 2022-01-27; First posted 2022-02-08 (Actual); Last update posted 2022-08-29 (Actual); Status verified 2022-08

CONDITIONS: Kidney Transplantation; Glomerular Filtration Rate
Keywords: Glomerular filtration rate; Kidney transplantation; Equation; Prediction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (8):
- Development cohort: kidney transplant recipients in 3 centres in France: Necker, Saint-Louis and Toulouse hospitals
  Interventions: Other: No intervention
- Validation cohort 1: kidney transplant recipients from Montpellier Hospital, France
  Interventions: Other: No intervention
- Validation cohort 2: kidney transplant recipients from Lyon Hospital, France
  Interventions: Other: No intervention
- Validation cohort 3: kidney transplant recipients from Tenon Hospital, France
  Interventions: Other: No intervention
- Validation cohort 4: kidney transplant recipients from Saint-Etienne Hospital, France
  Interventions: Other: No intervention
- Validation cohort 5: kidney transplant recipients from Mayo Clinic Hospital, USA
  Interventions: Other: No intervention
- Validation cohort 6: kidney transplant recipients from Bergamo hospital, Italy
  Interventions: Other: No intervention
- Validation cohort 7: kidney transplant recipients from Zagreb hospital, Croatia
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Kidney recipients aged over 18 and of all sexes recruited from 2000 who have mGFR follow-up and clinical, biological, and immunological data

SUMMARY:
Accurate estimation of the glomerular filtration rate (GFR) is crucial for the management of kidney recipients, since it is the most predictive parameter of allograft failure that drives patient monitoring and decision-making. Standard and recent race-free GFR equations have been developed in native kidneys, but their performances in transplant kidney population remains unknown. We aimed at developing a kidney-transplant-specific GFR equation, and comparing its performance to standard GFR equations.

DETAILED DESCRIPTION:
Historically, GFR equations, which predict the measured GFR (mGFR), were developed on patients with native kidneys and were further validated and used in kidney recipients. However, studies have shown significant heterogeneity in the performances of GFR equations when applied in kidney recipients, which may be attributed to variations and intrinsic characteristics specific to the transplant population. We thus made the hypothesis that GFR equations developed on a large, well-phenotyped kidney recipient cohort might achieve good performances in predicting mGFR.

The project therefore aims to:

1. Develop new kidney-recipient-specific (KRS) GFR equations and compare their performances with the standard GFR equations
2. Investigate whether the use of race increasers the performances of the new kidney-recipient-specific (KRS) GFR equations
3. Evaluate the effects of the new equations on the chronic kidney disease (CKD) prevalence and GFR stage

This study will provide us with data of kidney transplant patients that may allow the development of a new KRS GFR equation.

A new KRS GFR equation that presents with increased performances, as compared to current GFR equations, will improve the GFR calculation in kidney recipients, and therefore improve clinical decisions and the long-term kidney allograft management. Decisions regarding the return to dialysis or placement on the transplant waiting list will be taken with more accuracy and therefore potentially improve the financial allocation of kidney transplantation for the society.

ELIGIBILITY:
Inclusion Criteria:

* Living or deceased donor kidney recipient transplanted between 01/01/2000 and 01/01/2021.
* Men or women over 18 years of age.
* Written informed consent at the time of transplantation for the center database.

Exclusion Criteria:

• Combined transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The development cohort consisted of kidney transplant recipients from 3 centres in France. The validation cohorts consisted kidney transplant recipients from 6 centers in Europe and 1 in the Unites states.
Sampling Method: Probability Sample
Enrollment: 11412 (Actual)
Dates: Start 2000-01-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Measured glomerular filtration rate (mGFR) | Up to 15 years after kidney transplantation
  Isotopic measurements of GFR

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Loupy, MD, PhD, Principal Investigator — Paris Translational Research Center for Organ Transplantation
Locations (10):
- William J. von Liebig Centre for Transplantation and Clinical Regeneration, Mayo Clinic, Rochester, Minnesota, United States
- Department of Nephrology, Arterial Hypertension, Dialysis and Transplantation, University Hospital Centre Zagreb, School of Medicine, University of Zagreb, Zagreb, Croatia
- France (7):
  - Department of Transplantation, Nephrology and Clinical Immunology, Hospices Civils de Lyon, Lyon
  - Department of Nephrology, Centre Hospitalier Universitaire, Montpellier, Montpellier
  - Kidney Transplant Department, Necker Hospital, Assistance Publique - Hôpitaux de Paris, Paris
  - Kidney Transplant Department, Saint-Louis Hospital, Assistance Publique - Hôpitaux de Paris, Paris
  - Kidney Transplant Department, Tenon Hospital, Assistance Publique - Hôpitaux de Paris, Paris
  - Nephrology, Dialysis and Renal Transplantation Department, Hôpital Nord, CHU de Saint-Etienne, Jean Monnet University, Université de Lyon, Saint-Etienne
  - Department of Nephrology and Organ Transplantation, CHU Rangueil, Toulouse
- Istituto di Ricerche Farmacologiche Mario Negri IRCCS, Bergamo, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Raynaud M, Al-Awadhi S, Juric I, Divard G, Lombardi Y, Basic-Jukic N, Aubert O, Dubourg L, Masson I, Mariat C, Prie D, Pernin V, Le Quintrec M, Larson TS, Stegall MD, Bikbov B, Ruggenenti P, Mesnard L, Ibrahim HN, Nielsen MB, Matas AJ, Nankivell BJ, Benjamens S, Pol RA, Bakker SJL, Jouven X, Legendre C, Kamar N, Smith BH, Wadei HM, Durrbach A, Vincenti F, Remuzzi G, Lefaucheur C, Bentall AJ, Loupy A. Race-free estimated glomerular filtration rate equation in kidney transplant recipients: development and validation study. BMJ. 2023 May 31;381:e073654. doi: 10.1136/bmj-2022-073654. PMID 37257905